CLINICAL TRIAL: NCT04649580
Title: A Cross-Sectional Patient-Reported Study To Assess The Patient Preference Of Treatment Administration Setting, Impact On Health-Related Quality Of Life, Work Productivity, Wider Societal Costs And Healthcare Utilisation For Patients With Gastroenteropancreatic Neuroendocrine Tumours (GEP-NETs) Prescribed Somatuline® Autogel® In A Homecare Setting and Hospital Setting.
Brief Title: United Kingdom (UK) Patient Preference Study of Somatuline Autogel and Treatment Administration Setting
Acronym: PREF-NET
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-GB-52030-394
Record Dates: First submitted 2020-09-23; First posted 2020-12-02 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Neuroendocrine Tumours (NET)
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Online Survey
- One-to-one interviews

SUMMARY:
The aim of the study is to generate real-world evidence to describe the patient experience of administration of Somatuline® Autogel® (lanreotide) in homecare and hospital settings, and the associated impact on healthcare utilisation, societal cost, work productivity and health-related quality of life (HRQoL)

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of GEP-NETs
* Patients on prescribed lanreotide Autogel®;
* Patients who have switched from hospital to homecare administration setting at least 2 months ago
* Patients judged to be on a stable dose; 120mg for tumour control or >1 injection at same dose for symptom control

Exclusion Criteria:

* Patients who decline or lack capacity to consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UK patients with NET receiving Somatuline Autogel injections at home
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Patient preferences of treatment administration setting (homecare or hospital) | Baseline
  Survey responses of patient experience of injections at home and compared to responses of patient experience of injections when given in hospital

SECONDARY OUTCOMES:
Demographic characteristics of enrolled patients with GEP-NETs | Baseline
  Age (years); Gender (male, female); Current employment status: full time, part time, unemployed, retired, student, homemaker, unpaid carer)
Clinical characteristics of enrolled patients with GEP-NETs | Baseline
  Disease duration; Duration of homecare administration of lanreotide; Duration of hospital administration of lanreotide
Patient-reported impact on healthcare resource use | Baseline
  Assessed using bespoke questionnaire a patient-reported opinion on how homecare administration compares to hospital administration (i.e. much worse / somewhat worse / about the same / somewhat better / much better) for the number of administration setting related aspects described in the protocol, as well as choosing the most applicable answer(s) where applicable.
Patient-reported impact on wider societal costs | Baseline
  Assessed using bespoke questionnaire a patient-reported opinion on how homecare administration compares to hospital administration (i.e. much worse / somewhat worse / about the same / somewhat better / much better) for the number of administration setting related aspects described in the protocol, as well as choosing the most applicable answer(s) where applicable.
Patient-reported work productivity | Baseline
  Assessed using the Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH) and bespoke questionaire
Description of patient-reported HRQoL | Baseline
  Assessed using bespoke questionnaire a patient-reported opinion on how homecare administration compares to hospital administration (i.e. much worse / somewhat worse / about the same / somewhat better / much better) for the number of administration setting related aspects described in the protocol, as well as choosing the most applicable answer(s) where applicable.)
Description of patient experience of taking lanreotide in the hospital and homecare settings and reported benefits/limitations of each setting; | 1 month
  Assessed using qualitative interviews which will be conducted over the telephone by an experienced qualitative interviewer. During the interview semi-structured interview guide will be used, based on guidance and feedback from a clinical expert (specialist nurse) and patient expert(s). The interviews will be primarily guided by the questions in the discussion guide; however, participants will be free to direct the conversation to topics they feel are relevant to their experience.
Description of the impact of the homecare and hospital settings on HRQoL, work productivity, emotional and physical health | 1 month
  Assessed using qualitative interviews which will be conducted over the telephone by an experienced qualitative interviewer. During the interview semi-structured interview guide will be used, based on guidance and feedback from a clinical expert (specialist nurse) and patient expert(s). The interviews will be primarily guided by the questions in the discussion guide; however, participants will be free to direct the conversation to topics they feel are relevant to their experience.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cardiff and Vale University LHB, Cardiff
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Royal Free London NHS Foundation Trust, London

REFERENCES:
- See also: Related Info — https://link.springer.com/article/10.1007/s00520-024-08377-7